CLINICAL TRIAL: NCT07314203
Title: Clinical Efficacy of Adebrelimab With or Without Apatinib Mesilate and SOX Neoadjuvant Therapy in Locally Advanced Gastric Cancer
Acronym: SOP-XH-IRB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Chief doctor, phD, FACS, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOP-XH-IRB
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Surgery
Keywords: gastric cancer; neoadjuvant therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research group (Experimental): Study population received the combination of Adabelimab, Apatinib Mesylate, and SOX regimen
  Interventions: Drug: Apatinib Mesylate Tablets

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — Apatinib Mesylate

SUMMARY:
Exploring the pathological complete response rate (pCR) of locally advanced gastric cancer treated with adebelimab combined or not combined with apatinib mesylate and SOX neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

**Inclusion Criteria** 1. Age 18-75 years (inclusive). 2. Histologically or cytologically confirmed unresectable, locally advanced or metastatic HER2-negative adenocarcinoma of the stomach or gastro-oesophageal junction (GEJ).

3. No prior systemic chemotherapy, radiotherapy, targeted therapy, or immunotherapy for advanced disease. Subjects who have received prior (neo)adjuvant chemotherapy and/or radiotherapy are eligible provided the last dose was completed ≥ 6 months before randomisation.

4. At least one measurable lesion per RECIST 1.1 (see Appendix 2). 5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1 (see Appendix 4).

6. Estimated life expectancy > 3 months. 7. Adequate major organ function defined as:

1. Haematology (obtained ≤ 14 days without transfusion):

   1. Hb ≥ 80 g/L
   2. WBC ≥ 3 × 10⁹/L
   3. ANC ≥ 1.5 × 10⁹/L
   4. PLT ≥ 100 × 10⁹/L
2. Biochemistry:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN)
   2. ALT and AST < 2.5 × ULN; ALP ≤ 1.5 × ULN
   3. Serum creatinine ≤ 1 × ULN and calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula) 8. Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to enrolment and must use highly effective contraception from screening until 8 weeks after the last dose of study drug. Men must be surgically sterile or agree to use effective contraception during the same period.

      9. No participation in any other interventional clinical trial during the pre-treatment or on-treatment phases of this study.

      10. Voluntary written informed consent obtained; willing and able to comply with study procedures and follow-up.

      Exclusion Criteria:

      Exclusion Criteria

      Subjects meeting any of the following conditions will be excluded from enrollment:
      1. Known or suspected hypersensitivity to the investigational drug or any drug of the same class.
      2. Other malignancies within the past 5 years, except adequately treated basal-cell or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix.
      3. Currently receiving treatment in another interventional clinical trial, or any systemic anti-gastric-cancer therapy within 4 weeks prior to the first dose.
      4. Systemic Chinese patent medicines with anti-tumor indications or immunomodulatory agents (e.g., thymosin, interferon, interleukins; local intrapleural use for effusion control is permitted) received within 2 weeks before the first dose.
      5. Prior exposure to: anti-PD-1, anti-PD-L1, anti-PD-L2, or any agent targeting other T-cell co-stimulatory or co-inhibitory pathways (including but not limited to CTLA-4, OX-40, CD137); or prior chemotherapy including S-1.
      6. Live-vaccine administration within 4 weeks before enrollment or planned during the study.

         Note: Inactivated seasonal influenza vaccine by injection is allowed within 4 weeks; intranasal live-attenuated influenza vaccine is prohibited.
      7. Active autoimmune disease requiring systemic therapy (e.g., immunosuppressants, corticosteroids, or disease-modifying agents) within 2 years before the first dose. Replacement therapy (thyroxine, insulin, physiologic glucocorticoids for adrenal or pituitary insufficiency) is not considered systemic therapy.
      8. Prior allogeneic bone-marrow or solid-organ transplantation.
      9. Any condition that could impair drug absorption or inability to swallow oral medication.
      10. Uncontrolled hypertension despite optimal medical management:

          * SBP ≥ 150 mmHg or DBP ≥ 100 mmHg on a single antihypertensive, or requirement of ≥ 2 antihypertensive agents.
      11. Urinalysis showing proteinuria ≥ 2+ and 24-h urinary protein > 1.0 g.
      12. Active gastro-duodenal ulcer, ulcerative colitis, or other gastrointestinal disorders with bleeding risk; un-resected tumors with active hemorrhage; or any other condition judged by the investigator to predispose to GI bleeding or perforation.
      13. Significant bleeding tendency within 3 months before enrollment: overt bleeding > 30 mL, hematemesis, melena, hematochezia; hemoptysis (> 5 mL fresh blood within 4 weeks); or thrombo-embolic event (including stroke/TIA) within 12 months.
      14. Clinically significant cardiovascular disease:

          * Acute MI, unstable/severe angina, or CABG within 6 months before enrollment;
          * NYHA class > II congestive heart failure;
          * Ventricular arrhythmia requiring therapy;
          * QTc ≥ 480 ms on baseline ECG.
      15. Active or uncontrolled severe infection (≥ CTCAE grade 2).
      16. Known HIV infection; clinically significant hepatic disorders:

          * Chronic hepatitis B with active replication (HBV DNA > 1 × 10⁴ copies/mL or > 2000 IU/mL);
          * Hepatitis C with detectable HCV RNA (> 1 × 10³ copies/mL);
          * Other hepatitis or cirrhosis.
      17. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
      18. Any condition that, in the opinion of the investigator, would compromise the subject's safety or interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Estimated)
Dates: Start 2026-12-25 (Estimated); Primary Completion 2027-08-25 (Estimated); Study Completion 2028-08-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 day
  Objective Response Rate (ORR) is defined as the proportion of patients with confirmed complete response (CR) or partial response (PR) based on standardized, objective criteria (e.g., RECIST 1.1).

SECONDARY OUTCOMES:
Median Overall Survival | according to the OS
  Median Overall Survival (OS) is defined as the time from the date of diagnosis or initiation of treatment to the point at which 50% of patients have died (or reached the study endpoint event), serving as a key indicator for evaluating treatment efficacy and prognosis in chronic diseases such as cancer.
Progression-Free Survival | 36 months
  Progression-Free Survival (PFS) is defined as the time from randomization (or initiation of treatment) to the first documented disease progression (PD) or death from any cause, whichever occurs first
Duration of Response | 1 day
  Duration of Response (DOR) is defined as the time from the first documented complete response (CR) or partial response (PR) until disease progression (PD) or death from any cause, whichever occurs first.
Adverse Event | 30 days
  Adverse Event (AE) Incidence Rate is defined as the proportion of participants in a defined analysis set who experience at least one adverse event during a specified observation period after initiation of an intervention (drug, device, or procedure); it quantifies the frequency of intervention-related risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No